CLINICAL TRIAL: NCT00478673
Title: The NexStent® Carotid Stent System: A Post Market Approval Evaluation Study In Conjunction With the FilterWire EZ™ Embolic Protection System
Brief Title: Post-Approval Study of the NexStent Carotid Stent System and the FilterWire EZ Embolic Protection System: SONOMA
Acronym: SONOMA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was terminated in June 2008 due to market withdrawal of the NexStent Carotid Stent System.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2042; SONOMA
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Carotid Stenosis
Keywords: NexStent; FilterWire EZ; Boston Scientific; Carotid Artery; Carotid Endarterectomy; Carotid Revascularization
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NexStent Carotid Stent System (Monorail Delivery System) — Self-expanding carotid stent for treating patients at high risk for adverse events from carotid endarterectomy who require carotid revascularization.
Device: FilterWire EZ™ Embolic Protection System — Used as a guide wire and embolic protection system to contain and remove embolic material (thrombus/debris) while performing angioplasty and stenting procedures in coronary saphenous vein bypass grafts and carotid arteries.

SUMMARY:
The primary objective of the SONOMA Registry is to confirm the safety of the NexStent® Carotid Stent System and FilterWire EZ™ Embolic Protection System in routine clinical practice and to identify rare or unanticipated device-related events that might occur.

DETAILED DESCRIPTION:
The SONOMA Registry will enroll approximately 300 subjects at a maximum at 78 study centers.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must be indicated for carotid stent placement as per NexStent Carotid Stent labeling located in the Directions for Use (DFU).

Exclusion Criteria:

* Subjects with contraindications as outlined in the DFU should be excluded from this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subbarao Myla, M.D., Principal Investigator — Hoag Memorial Hospital; Pamela Grady, PhD, Study Director — Boston Scientific Corporation
Locations (62):
- United States (62):
  - Huntsville Hospital Heart Center, Huntsville, Alabama
  - St. Luke's Medical Center, Phoenix, Arizona
  - Central Cardiology Medical Clinic, Bakersfield, California
  - Los Angeles Cardiology Associates, Los Angeles, California
  - ACS Research Group, Inc., Mountain View, California
  - Hoag Memorial Hospital / Presbyterian, Newport Beach, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - JFK Medical Center, Atlantis, Florida
  - Northwest Medical Center, Margate, Florida
  - Baptist Cardiac and Vascular Institute, Baptist Hospital of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Neurological Institute of Savannah, Savannah, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis Knighton Medical Center, Shreveport, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Great Lakes Heart & Vascular Institute, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Michigan Heart PC, Ypsilanti, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - St. Anthony's Medical Center, St Louis, Missouri
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial, Morristown, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Kaleida Health, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Buffalo Neurosurgery Group, Williamsville, New York
  - Cleveland Clinic and Foundation, Cleveland, Ohio
  - Ohio State University Medical, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Heritage Valley Health System, Beaver, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Center PA Cardiovascular Research Institute, Harrisburg, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - St. Mary Medical Center, Yardley, Pennsylvania
  - York Hospital, York, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Cardiovascular Associates, PC Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Dallas Fort Worth Vascular, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Central Cardiovaascular Research Foundation, San Antonio, Texas
  - Washington Cardiovscular Research and Education Foundation, Seattle, Washington
  - St. Joseph Regional Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Qureshi AI, Knape C, Maroney J, Suri MF, Hopkins LN. Multicenter clinical trial of the NexStent coiled sheet stent in the treatment of extracranial carotid artery stenosis: immediate results and late clinical outcomes. J Neurosurg. 2003 Aug;99(2):264-70. doi: 10.3171/jns.2003.99.2.0264. PMID 12924698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on May 23, 2007. Enrollment was suspended on June 6, 2008, due to a voluntary recall of the NexStent Carotid Stent System. On June 17, 2008, enrollment was terminated and the NexStent Carotid Stent System was withdrawn from the market.
Groups:
- NexStent Carotid Stent System: Subjects in this arm had carotid artery disease treated with the NexStent Carotid Stent System used in conjunction with the FilterWire EZ Embolic Protection System. The NexStent Carotid Stent is a rolled metal mesh sheet constrained in a sheath. The stent is inserted through the groin and is opened in the blocked carotid artery. The FilterWire EZ Embolic Protection System is a temporary filtration system used to contain and remove embolic material that may be released during the stenting procedure.
Period: 30-Days Post-Procedure
Arm/Group | NexStent Carotid Stent System
Started | 298
Completed | 288 (7 participants who did not complete this Period due to "Missed Visit" still continued on to Period 2)
Not Completed | 10
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Missed Visit | 7
Period: 12-Months Post-Procedure
Arm/Group | NexStent Carotid Stent System
Started | 295 (3 participants who did not complete Period 1 due to death (2) and withdrawal (1) are not included.)
Completed | 231
Not Completed | 64
Not completed — Death | 23
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 6
Not completed — Missed Visit | 25
Not completed — Visit Not Required by Protocol | 6

BASELINE CHARACTERISTICS:
Arm/Group | NexStent Carotid Stent System
Number analyzed (Participants) | 298
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 179
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 15
  Caucasian | 258
  Asian | 2
  Black, of African Heritage | 20
  Native Hawaiian or Other Pacific Islander | 0
  American Indian or Alaska Native | 1
  Other | 2
Region of Enrollment [Number; unit: Participants]
  United States | 298
Current Carotid Bruit [Number; unit: Participants]
  Current Carotid Bruit | 175
  No Current Carotid Bruit | 82
  Unknown | 41
History of Carotid Atherosclerosis [Number; unit: Participants]
  History of Carotid Atherosclerosis | 187
  No History of Carotid Atherosclerosis | 101
  Unknown | 10
History of Transient Ischemic Attack (TIA) [Number; unit: Participants]
  History of TIA | 77
  No History of TIA | 207
  Unknown | 14
History of Cerebrovascular Accident (CVA) [Number; unit: Participants]
  History of CVA | 62
  No History of CVA | 233
  Unknown | 3
History of Vertebrobasilar Occlusive Disease [Number; unit: Participants]
  History of Vertebrobasilar Occlusive Disease | 11
  No History of Vertebrobasilar Occlusive Disease | 267
  Unknown | 20
History of Seizure [Number; unit: Participants]
  History of Seizure | 5
  No History of Seizure | 290
  Unknown | 3
History of Carotid Endarterectomy (CEA) [Number; unit: Participants]
  History of CEA | 74
  No History of CEA | 223
  Unknown | 1
History of Percutaneous Transluminal Angioplasty (PTA) [Number; unit: Participants]
  History of PTA | 15
  No History of PTA | 282
  Unknown | 1
History of Carotid Restenosis [Number; unit: Participants]
  History of Carotid Restenosis | 49
  No History of Carotid Restenosis | 246
  Unknown | 3
History of Upper Extremity Fibromuscular Dysplasia (FMD) [Number; unit: Participants]
  History of Upper Extremity FMD | 1
  No History of Upper Extremity FMD | 292
  Unknown | 5
History of Coronary Artery Disease (CAD) [Number; unit: Participants]
  History of CAD | 196
  No History of CAD | 94
  Unknown | 8
History of Myocardial Infarction (MI) [Number; unit: Participants]
  History of MI | 81
  No History of MI | 206
  Unknown | 11
History of Congestive Heart Failure (CHF) [Number; unit: Participants]
  History of CHF | 54
  No History of CHF | 241
  Unknown | 3
Current Angina [Number; unit: Participants]
  Stable Angina | 42
  Unstable Angina | 10
  Silent Ischemia | 3
  None | 243
History of Percutaneous Coronary Intervention (PCI) [Number; unit: Participants]
  History of PCI | 97
  No History of PCI | 196
  Unknown | 5
History of Coronary Artery Bypass Grafting (CABG) [Number; unit: Participants]
  History of CABG | 85
  No History of CABG | 212
  Unknown | 1
History of Atrial Fibrillation/Flutter [Number; unit: Participants]
  History of Atrial Fibrillation/Flutter | 50
  No History of Atrial Fibrillation/Flutter | 241
  Unknown | 7
History of Smoking [Number; unit: Participants]
  Current | 67
  Previous | 145
  Never | 77
  Unknown | 9
History of Diabetes [Number; unit: Participants]
  History of Diabetes | 114
  No History of Diabetes | 182
  Unknown | 2
History of Hyperlipidemia [Number; unit: Participants]
  History of Hyperlipidemia | 257
  No History of Hyperlipidemia | 40
  Unknown | 1
History of Hypertension [Number; unit: Participants]
  History of Hypertension | 268
  No History of Hypertension | 29
  Unknown | 1
History of Peripheral Vascular Disease (PVD) [Number; unit: Participants]
  History of PVD | 117
  No History of PVD | 172
  Unknown | 9
History of Significant Bleeding [Number; unit: Participants]
  History of Significant Bleeding | 11
  No History of Significant Bleeding | 286
  Unknown | 1
History of Mantle or Head and Neck Radiation [Number; unit: Participants]
  History of Mantle or Head and Neck Radiation | 15
  No History of Mantle or Head and Neck Radiation | 281
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a 30-Day Major Adverse Event (MAE)
Description: 30-day major adverse events (MAEs) are defined as all deaths, strokes, and myocardial infarctions (MIs) that occur within 0-30 days post-procedure.
Time Frame: 30 Days
Population: ITT Analysis: All enrolled subjects who experienced a 30-day MAE and/or completed a follow-up evaluation >=23 days post-procedure were evaluable. Subjects who experienced more than one MAE within 30 days were counted in the number of subjects with each applicable event, but were only counted once in the number of subjects with overall 30-day MAE.
Measure: Number; unit: Participants
Arm/Group | NexStent Carotid Stent System
Number analyzed (Participants) | 293
Participants
  30-Day Major Adverse Events (Overall) | 13
  Death (0-30 Days) | 3 [2.4 to 7.5]
  Stroke (0-30 Days) | 10
  MI (0-30 Days) | 3

2. Primary Outcome: Number of Participants Who Experienced a 12-Month Major Adverse Event (MAE)
Description: 12-month major adverse events (MAEs) are defined as all deaths, strokes, and myocardial infarctions (MIs) that occur within 0-30 days post-procedure (see 30-Day MAE above), and ipsilateral stroke events that occur within 31-365 days post-procedure.
Time Frame: 12 Months
Population: ITT Analysis: All enrolled subjects who experienced a 12-mo MAE and/or completed a follow-up evaluation >=335 days post-procedure were evaluable. Subjects who experienced more than one MAE within 12 months were counted in the number of subjects with each applicable event, but were only counted once in the number of subjects with overall 12-mo MAE.
Measure: Number; unit: Participants
Arm/Group | NexStent Carotid Stent System
Number analyzed (Participants) | 235
Participants
  12-Month Major Adverse Events (Overall) | 16
  Ipsilateral Stroke (31-365 Days) | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the 12-month follow-up evaluation. Data reported here represent the total study experience.
Description: Subjects were evaluated for adverse events during the procedure, at hospital discharge and at each follow-up visit.
Arm/Group | NexStent Carotid Stent System
Serious Adverse Events (participants affected / at risk) | 150/298
Other Adverse Events (participants affected / at risk) | 72/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NexStent Carotid Stent System (N=298)
Anaemia (Blood and lymphatic system disorders) | 14 (14)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 7 (11)
Atrial fibrillation (Cardiac disorders) | 7 (8)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 6 (6)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 12 (18)
Coronary artery disease (Cardiac disorders) | 3 (3)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 8 (10)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blindness transient (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (3)
Asthenia (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 12 (13)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Chest wall abscess (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Post procedural infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 5 (5)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Cephalhaematoma (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 4 (4)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (2)
Carotid artery dissection (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 16 (18)
Carotid artery thrombosis (Nervous system disorders) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 7 (7)
Convulsion (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Intention tremor (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Postictal paralysis (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 8 (8)
Conversion disorder (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 5 (6)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Renal hypertension (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 3 (3)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 20 (20)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (5)
Peripheral vascular disorder (Vascular disorders) | 3 (4)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NexStent Carotid Stent System (N=298)
Carotid artery stenosis (Nervous system disorders) | 53 (54)
Hypotension (Vascular disorders) | 24 (26)

LIMITATIONS AND CAVEATS:
Enrollment was terminated in June 2008 due to market withdrawal of the NexStent Carotid Stent System. The early termination of enrollment led to a smaller than expected number of analyzable subjects (298 actual vs. 1500 anticipated).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication to remove any confidential information or other proprietary information of Sponsor.